CLINICAL TRIAL: NCT01918254
Title: Phase IB, Open-Label, Multicenter, Dose-Escalation Study Followed by an Extension Phase to Evaluate the Safety, Pharmacokinetics and Activity of RO5479599, a Glycoengineered Antibody Against HER3, Administered in Combination With Pertuzumab and Paclitaxel in Patients With Metastatic Breast Cancer Expressing HER3 & HER2 Protein
Brief Title: A Study to Evaluate Lumretuzumab in Combination With Pertuzumab and Paclitaxel in Participants With Metastatic Breast Cancer Expressing Human Epidermal Growth Factor Receptor (HER) 3 and HER2 Protein
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BP28752; 2013-000090-67 (EudraCT Number)
Record Dates: First submitted 2013-07-03; First posted 2013-08-07 (Estimated); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel; pertuzumab; lumretuzumab

ARMS (3):
- Lumretuzumab Dose Escalation (Experimental): Participants will receive escalating doses of lumretuzumab starting at 1000 mg IV (on Day 1, except Cycle 1 where lumretuzumab will be administered on Day 2) along with paclitaxel 80 mg/m^2 IV (on Days 1, 8, and 15), and pertuzumab 840 mg IV (on Day 1) initial dose followed by 420 mg IV, in each 21-day cycle. Participants will be treated until disease progression, unacceptable toxicities, and withdrawal from treatment for other reasons or death.
  Interventions: Drug: Paclitaxel; Drug: Pertuzumab; Drug: Lumretuzumab
- EPC1: Lumretuzumab (Prior Chemotherapy) (Experimental): Extension phase Cohort 1 (EPC1): Participants will receive lumretuzumab 1000 mg IV (on Day 1) along with paclitaxel 80 mg/m^2 IV (on Days 1, 8, and 15), and pertuzumab 840 mg IV (on Day 1) initial dose followed by 420 mg IV, in each 21-day cycle. Participants will be treated until disease progression, unacceptable toxicities, and withdrawal from treatment for other reasons or death.
  Interventions: Drug: Paclitaxel; Drug: Pertuzumab; Drug: Lumretuzumab
- EPC2: Lumretuzumab (Without Prior Chemotherapy) (Experimental): Extension phase Cohort 2 (EPC2): Participants will receive lumretuzumab 2000 mg IV (on Day 1) along with paclitaxel 80 mg/m^2 IV (on Days 1, 8, and 15), and pertuzumab 420 mg IV (on Day 1), in each 21-day cycle. Participants will be treated until disease progression, unacceptable toxicities, and withdrawal from treatment for other reasons or death. Only participants with no prior chemotherapy for metastatic disease and/or a maximum of only one prior chemotherapy regimen in adjuvant or neoadjuvant setting will be enrolled in this cohort.
  Interventions: Drug: Paclitaxel; Drug: Pertuzumab; Drug: Lumretuzumab

INTERVENTIONS:
Drug: Paclitaxel — Paclitaxel IV infusion will be administered as per schedule described in individual arm.
Drug: Pertuzumab — Pertuzumab IV infusion will be administered as per schedule described in individual arm.
  Other Names: Perjeta
Drug: Lumretuzumab — Lumretuzumab will be administered as per schedule described in individual arm.
  Other Names: RO5479599; RG7116

SUMMARY:
This multicenter, open-label dose-escalation study with an extension phase will evaluate the safety and pharmacokinetics of lumretuzumab in combination with pertuzumab and paclitaxel in participants with metastatic breast cancer expressing HER3 and HER2 protein. Cohorts of participants will receive escalating doses of lumretuzumab intravenously (IV) every three weeks (Q3W) in combination with pertuzumab 840 milligrams (mg) IV initial dose followed by 420 mg IV Q3W and paclitaxel 80 milligrams per square meter (mg/m^2) IV weekly. After completion of dose-limiting toxicity period (21 days), the study will be conducted in two extension phase cohorts: Cohort 1 and Cohort 2. Enrollment in Extension Phase Cohort 2 will occur only upon completion of Extension Phase Cohort 1. Anticipated time on study treatment is until disease progression or unacceptable toxicity occurs.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic breast cancer expressing HER3 and HER2 protein
* Participants must be willing to undergo a fresh (pretreatment) tumor/metastases biopsy that will be used to assess the level of HER3 protein expression by immunohistochemistry (IHC) and central pathology review
* HER2 status confirmed on same tumor/metastases by a central laboratory. Breast cancer tumors and/or metastases must be HER2 IHC 1+/in-situ hybridization (ISH)- or HER2 ICH 2+/ISH- as assessed by parallel testing of protein and gene amplification using a Food and Drug Administration (FDA)-approved test
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1
* Taxane-naive participants or participants who have received taxanes as part of an adjuvant/neoadjuvant treatment regimen with a disease-free interval of at least 1 year. Participants who have received a docetaxel-containing regimen in the metastatic setting may be eligible. Participants who have received paclitaxel/nab-paclitaxel in the metastatic setting but have discontinued paclitaxel/nab-paclitaxel for a reason other than disease progression and have had a taxane-free interval of at least 6 months may be eligible unless otherwise contraindicated at the investigator's discretion
* Radiologically measurable or clinically evaluable disease according to RECIST criteria
* Last dose of systemic anti-neoplastic therapy greater than (>) 21 days prior to first study treatment infusion. Palliative radiotherapy is allowed up to 2 weeks before the first study treatment infusion
* All acute toxic effects of any prior radiotherapy, chemotherapy or surgical procedure must have resolved to Grade less than or equal to (<=) 1, except alopecia (any grade)
* Adequate hematological, liver and renal function
* Baseline left ventricular ejection fraction (LVEF) of greater than or equal to (>=) 50 percent (%) (measured by echocardiography)
* Female participants of childbearing potential and male participants must agree to use effective contraception as defined by protocol during the study and for at least 6 months after the last dose of study medication
* Participants with Gilbert's Syndrome will be eligible for the study

For extension Phase 2, all of the above except the inclusion criteria mentioned for taxane-naive participants or participants who have received taxanes. In addition, participants in extension Phase 2 may include:

* Participants with no prior chemotherapy for metastatic breast cancer and/or a maximum of only one prior chemotherapy regimen in the adjuvant or neoadjuvant setting
* Taxane-naive participants or participants who have received taxanes as a part of an adjuvant/neoadjuvant treatment regimen with a disease-free interval of at least 1 year

Exclusion Criteria:

* History of clinical evidence of central nervous system (CNS) primary tumors or metastases including leptomeningeal metastases unless they have been previously treated, are asymptomatic and have had no requirement for steroids or enzyme-inducing anti-convulsants in the last 14 days
* Evidence of significant, uncontrolled concomitant diseases which could affect compliance with the protocol or interpretation of results, including uncontrolled diabetes mellitus
* Active or uncontrolled infections
* Known human immunodeficiency virus (HIV) or known active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection
* Major surgery or significant traumatic injury less than (<) 28 days prior to first study treatment infusion (excluding biopsies) or anticipation of the need for a major surgery during study treatment
* Pregnant or breast-feeding women
* Known hypersensitivity to any of the components of RO5479599, pertuzumab or paclitaxel
* Participants with contraindications for paclitaxel therapy according to the Summary of Product Characteristics (SmPC)
* Therapy with an antibody or immunotherapy concurrently or within a period of time where drug exposure is still considered biologically active (usually <5 times t1/2) prior to first dose of study treatment
* Regular immunosuppressive therapy (that is, for organ transplantation, chronic rheumatologic disease)
* Concurrent high doses of systemic corticosteroids (>20 milligrams [mg] of dexamethasone a day or equivalent for >7 consecutive days)
* Baseline QTc interval of >470 milliseconds (ms), participants with baseline resting bradycardia <45 beats per minute or baseline resting tachycardia >100 beats per minute
* Uncontrolled hypertension, unstable angina, congestive heart failure of any New York Heart Association (NYHA) classification, serious cardiac arrhythmia requiring treatment (exceptions: atrial fibrillation, paroxysmal supraventricular tachycardia), history of myocardial infraction within 6 months of enrollment or symptomatic LVEF dysfunction
* A history of Grade >=3 peripheral neuropathy of any etiology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2013-08-06 (Actual); Primary Completion 2016-10-07 (Actual); Study Completion 2016-10-07 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Dose-Limiting Toxicities (DLTs) | Day 1 up to Day 21
Percentage of Participants With Adverse Events | Baseline up to approximately 39 months
Percentage of Participants With Anti-Human Antibodies (HAHAs) to lumretuzumab [RO5479599] | Pre-infusion (Pr-I) (0 hour [h]) on Day 1 (D1) of each Cycle (Cy) up to approximately 39 months (assessed at Pr-I on D1 of each treatment Cy up to 28 and 42-45 days after last infusion [up to approximately 39 months overall]) (1 Cy = 21 days)
Pharmacokinetics: Area Under the Concentration-Time Curve (AUC) of lumretuzumab [RO5479599] | Pr-I (0 Hr) & 3, 24, 72, 168, 264, 312, 432, & 480 Hr post D1 infusion (infusion duration = 1.5-2 hours) of Cy4, 8 & post D2 infusion of Cy1; D1 of all other cycles up to 28 and 42-45 days after last dose (up to approximately 39 months) (1 Cy = 21 days)
Pharmacokinetics: Maximum Serum Concentration (Cmax) of lumretuzumab [RO5479599] | Pr-I (0 Hr) & 3, 24, 72, 168, 264, 312, 432, & 480 Hr post D1 infusion (infusion duration = 1.5-2 hours) of Cy4, 8 & post D2 infusion of Cy1; D1 of all other cycles up to 28 and 42-45 days after last dose (up to approximately 39 months) (1 Cy = 21 days)
Pharmacokinetics: Trough Serum Concentration (Ct) of lumretuzumab [RO5479599] | Pr-I (0 h) on D1 of each cycles beginning from Cy 2 up to 28 and 42-45 days after last infusion (up to approximately 39 months) (1 Cy = 21 days)
Pharmacokinetics: Time to Reach Maximum Serum Concentration (tmax) of lumretuzumab [RO5479599] | Pr-I (0 h) & 3, 24, 72, 168, 264, 312, 432, & 480 Hr post D1 infusion (infusion duration = 1.5-2 h) of Cy4, 8 & post D2 infusion of Cy1; D1 of all other cycles up to 28 and 42-45 days after last dose (up to approximately 39 months) (1 Cy = 21 days)
Pharmacokinetics: Clearance (CL) of lumretuzumab [RO5479599] | Pr-I (0 h) & 3, 24, 72, 168, 264, 312, 432, & 480 h post D1 infusion (infusion duration = 1.5-2 h) of Cy4, 8 & post D2 infusion of Cy1; D1 of all other cycles up to 28 and 42-45 days after last dose (up to approximately 39 months) (1 Cy = 21 days)
Pharmacokinetics: Volume of distribution (V) of lumretuzumab [RO5479599] | Pr-I (0 h) & 3, 24, 72, 168, 264, 312, 432, & 480 h post D1 infusion (infusion duration = 1.5-2 h) of Cy4, 8 & post D2 infusion of Cy1; D1 of all other cycles up to 28 and 42-45 days after last dose (up to approximately 39 months) (1 Cy = 21 days)
Pharmacokinetics: Accumulation Ratio of lumretuzumab [RO5479599] | Pr-I (0 h) & 3, 24, 72, 168, 264, 312, 432, & 480 h post D1 infusion (infusion duration = 1.5-2 h) of Cy4, 8 & post D2 infusion of Cy1; D1 of all other cycles up to 28 and 42-45 days after last dose (up to approximately 39 months) (1 Cy = 21 days)
Pharmacokinetics: Elimination Half-Life (t1/2) of lumretuzumab [RO5479599] | Pr-I (0 h) & 3, 24, 72, 168, 264, 312, 432, & 480 h post D1 infusion (infusion duration = 1.5-2 h) of Cy4, 8 & post D2 infusion of Cy1; D1 of all other cycles up to 28 and 42-45 days after last dose (up to approximately 39 months) (1 Cy = 21 days)
Pharmacokinetics: Serum Concentration at the Time of Tumor Progression (Cprog) of lumretuzumab [RO5479599] | At the time of tumor progression (up to approximately 39 months)
Pharmacokinetics: Serum Concentration at the Time of Tumor Response (Complete response [CR]/Partial Response [PR]) of lumretuzumab [RO5479599] | At the time of tumor progression (up to approximately 39 months)
Pharmacokinetics: Serum Concentration at the Time of DLT of lumretuzumab [RO5479599] | At the time of DLT (up to 21 days)
Pharmacokinetics: Serum Concentration at the Time of Tumor and Skin Biopsy (Cb) of lumretuzumab [RO5479599] | At the time of tumor/skin biopsy (up to approximately 39 months)
Pharmacokinetics: Serum Concentration at the Time of Infusion-Related Reactions (IRR) of lumretuzumab [RO5479599] | At the time of IRR (up to approximately 39 months)
Recommended Phase II Dose of lumretuzumab [RO5479599] | Day 1 up to Day 21

SECONDARY OUTCOMES:
Percentage of Participants With Best Overall Response of CR or PR (Objective Response) Assessed Using Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST V1.1) Criteria | Baseline up to documented disease progression (PD) or death, whichever occurs first up to approximately 39 months (assessed at baseline thereafter every 9 weeks up to 28 days after last infusion or early discontinuation)
Percentage of Participants With Best Overall Response of CR or PR or SD (Disease Control), Assessed Using RECIST V1.1 Criteria | Baseline up to documented PD or death, whichever occurs first up to approximately 39 months (assessed at baseline thereafter every 9 weeks up to 28 days after last infusion or early discontinuation)
Duration of Response, Assessed Using RECIST V1.1 Criteria | From first confirmed documented objective response (CR/PR) up to documented PD or death, whichever occurs first up to approximately 39 months (assessed at baseline thereafter every 9 weeks up to 28 days after last infusion or early discontinuation)
Progression-Free Survival Assessed Using RECIST V1.1 Criteria | Baseline up to documented PD or death, whichever occurs first up to approximately 39 months (assessed at baseline thereafter every 9 weeks up to 28 days after last infusion or early discontinuation)
Overall Survival | Baseline up to death (up to approximately 39 months)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (13):
- Rigshospitalet, Onkologisk Klinik, København Ø, Denmark
- France (4):
  - Centre Francois Baclesse; Comite Sein, Caen
  - Institut régional du Cancer Montpellier, Montpellier
  - Institut Curie; Oncologie Medicale, Paris
  - Institut Universitaire du Cancer - Oncopole Toulouse (IUCT-O), Toulouse
- Germany (3):
  - Universitaetsklinikum Essen; Westdeutsches Tumorzentrum; Innere Klinik (Tumorforschung), Essen
  - University of Hannover; Medical School, Hanover
  - Nationales Centrum für Tumorerkrankungen (NCT) ; Gyn. Onk. Frauenklinik; Uniklinikum Heidelberg, Heidelberg
- Spain (5):
  - Hospital del Mar; Servicio de Oncologia, Barcelona
  - Hospital Univ Vall d'Hebron; Servicio de Oncologia, Barcelona
  - Hospital Universitario 12 de Octubre; Servicio de Oncologia, Madrid
  - Centro Integral Oncologico Clara Campal (CIOCC); Dirección Médica, Madrid
  - Hospital Clinico Universitario de Valencia; Servicio de Onco-hematologia, Valencia

REFERENCES:
- [Derived] Schneeweiss A, Park-Simon TW, Albanell J, Lassen U, Cortes J, Dieras V, May M, Schindler C, Marme F, Cejalvo JM, Martinez-Garcia M, Gonzalez I, Lopez-Martin J, Welt A, Levy C, Joly F, Michielin F, Jacob W, Adessi C, Moisan A, Meneses-Lorente G, Racek T, James I, Ceppi M, Hasmann M, Weisser M, Cervantes A. Phase Ib study evaluating safety and clinical activity of the anti-HER3 antibody lumretuzumab combined with the anti-HER2 antibody pertuzumab and paclitaxel in HER3-positive, HER2-low metastatic breast cancer. Invest New Drugs. 2018 Oct;36(5):848-859. doi: 10.1007/s10637-018-0562-4. Epub 2018 Jan 19. PMID 29349598